CLINICAL TRIAL: NCT06776237
Title: Point of Care Ultrasound (PoCUS) as a Tool to Evaluate Patients at High Risk of Obstructive Sleep Apnea in the Obstetric Population
Brief Title: Point of Care Ultrasound in Pregnant Women (PoCUS-OB)
Status: Not yet recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Associate Professor, University Health Network, Toronto
Other Study IDs: 23-5451
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: OSA,Pregnancy,Women,HST,Ultrasound
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PoCUS — Participants after getting recruited will be asked for an ultrasonography of the neck. It will take around 30 minutes. At home, participants will be asked to wear a portable sleep study device overnight, to perform home sleep study. Although these devices are noninvasive and safe, they are not routinely used as a standard of care in the pregnant patient population.

SUMMARY:
Pregnant women with gestational age more than 20 weeks are at risk of developing Obstructive Sleep Apnea (OSA). OSA is a common underdiagnosed comorbid condition in pregnant women associated with adverse maternal and fetal outcomes. It is a severe form of sleep-disordered breathing (SDB), featured with repeated episodes of airflow reduction or cessation during sleep. It exists in different severity among pregnant women and maybe worsen over the course of the pregnancy. If OSA remains untreated, it can complicate the pregnancy by developing heart failure, gestational diabetes, pre-eclampsia, eclampsia, and hypertension. To determine the OSA during pregnancy has become an important issue to reduce the morbidity related to it. Currently, Polysomnography (PSG) remains the gold standard for diagnosing OSA, but scheduling and logistics remain significant impediments to accessibility for pregnant women. Home sleep apnea tests (HST) is a promising alternative but are expensive and not widely available. Point of care ultrasonography (PoCUS) is being increasingly used across specialties. Our preliminary data support the feasibility of PoCUS in the preoperative setting and increasing the diagnostic accuracy and the specificity for moderate to severe OSA (AHI >15 events per h) when combined with the STOP-Bang questionnaire (cut-off >5). Given that HST shows high levels of agreement with PSG for the diagnosis of OSA and are significantly less burdensome than PSG, investigators will evaluate the PoCUS airway examination against the HST for the diagnosis of OSA in pregnant women at high risk of OSA.

DETAILED DESCRIPTION:
This project is to define the range of mouth and tongue dimensions and to visualize airway structures by using ultrasound. Given that Home sleep apnea tests (HST) shows high levels of accuracy for the diagnosis of Obstructive sleep apnea (OSA), investigators hypothesize that the Point of care ultrasonography (PoCUS) airway examination against the HST for the diagnosis of OSA in pregnant women at the high-risk can,

1. reliably visualize upper airway structures that are responsible for OSA;
2. objectively measure airway soft tissue thickness and dimensions; and
3. identify pregnant women with moderate-severe OSA.

ELIGIBILITY:
- Inclusion criteria

* Pregnant women ≥ 18 years of age
* at > 20 weeks of gestation
* ASA physical status I - IV
* With untreated recently diagnosed (within the previous 12 months) OSA or at high risk of OSA will be eligible for inclusion.

High risk of OSA will be defined as outlined by Facco et al. and recommended by recently updated guidelines (i.e., score ≥ 75) (8).

- Exclusion criteria i) past history of oral, head or neck surgery (e.g., corrective surgery for OSA) ii) active head and neck disease (e.g., cancer, infection, radiotherapy etc.) iii) inability to perform HST per instruction iv) patients with diagnosed OSA on CPAP therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women ≥ 18 years of age
Study Population: Investigators aim to recruit 100 pregnant women ≥ 18 years of age at > 20 weeks of gestation, ASA physical status I - IV, with untreated recently diagnosed (within the previous 12 months) OSA or at high risk of OSA
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Areas Under the Curve (AUC) | One Day
  The primary outcome will be the difference in Areas Under the Curve (AUC) for each US parameter compared to the AUC of the HST obtained using the Receiver Operating Characteristic (ROC) curves for moderate to severe OSA defined as AHI > 15.

SECONDARY OUTCOMES:
The inter-rater reliability for measuring each one of the airway parameters | One Day
  i) The inter-rater reliability for measuring each one of the airway parameters ii) The association between each US parameter and OSA severity level (none/mild/moderate/severe) iii) The association between each US parameter and OSA diagnosis derived from PSG

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital (TWH)-University Health Network (UHN), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No